CLINICAL TRIAL: NCT01893294
Title: Phase I Trial of Intra-tumoral Gemcitabine Therapy for Locally Advanced Pancreatic Carcinoma
Brief Title: Gemcitabine Hydrochloride in Treating Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1241; NCI-2013-00798 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1241 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2015-10

CONDITIONS: Duct Cell Adenocarcinoma of the Pancreas; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Fluorouracil; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gemcitabine hydrochloride) (Experimental): Patients receive gemcitabine hydrochloride IT on day 1. Within 33 hours, patients receive standard chemotherapy comprising fluorouracil IV on days 1, 8, 15, 22, 29, and 36 and undergo standard radiation therapy 5 days a week for 6 weeks.
  Interventions: Drug: gemcitabine hydrochloride; Drug: fluorouracil; Radiation: radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IT
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of gemcitabine hydrochloride in treating patients with locally advanced pancreatic cancer. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerate dose (MTD) of intra-tumoral injection of gemcitabine (gemcitabine hydrochloride) when administered as a one time initial induction therapy in conjunction (=< 33 hours) prior to conventional multimodality treatment for locally advanced pancreatic cancer (LAPC).

SECONDARY OBJECTIVES:

I. To evaluate the initial and delayed toxicity associated with this treatment regimen.

OUTLINE: This is a dose-escalation study.

Patients receive gemcitabine hydrochloride intratumorally (IT) on day 1. Within 33 hours, patients receive standard chemotherapy comprising fluorouracil intravenously (IV) on days 1, 8, 15, 22, 29, and 36 and undergo standard radiation therapy 5 days a week for 6 weeks.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytology proven pancreatic ductal carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0,1 or 2
* Absolute neutrophil count (ANC) >= 1500
* Platelets (PLT) >= 100,000
* Hemoglobin (HgB) > 9.0 g/dL
* Total bilirubin < 2.0 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 5 x ULN
* Creatinine =< 1.5 mg/dL
* Negative pregnancy test done =< 14 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Imaging, a combination of at least two of the following (computed tomography [CT], magnetic resonance imaging [MRI], endoscopic ultrasound [EUS]) staging the pancreatic mass as "locally advanced"
* EUS clinically indicated for staging, and/or celiac neurolysis
* Resection declined by surgical staff based on designation of LAPC
* Willing to provide blood samples
* Willing to receive their standard multimodality therapy at Mayo Clinic, Rochester
* Willing to return to Mayo Clinic, Rochester during the observation phase

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Any prior treatment (chemotherapy, radiation) for pancreatic cancer
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 168 days (6 months), or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Prior pancreatic surgery
* Pancreatic tumor histology other than carcinoma (e.g. islet cell, lymphoma, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2015-10-30 (Actual)

PRIMARY OUTCOMES:
MTD of gemcitabine hydrochloride defined as the dose at which no more than 3 of 6 patients experience grade 3 or greater adverse events, as graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 4 weeks

SECONDARY OUTCOMES:
Incidence of immediate adverse events associated with this treatment, graded according to the NCI CTCAE version (v)3.0 | Within 72 hours of EUS
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Incidence of delayed adverse events associated with this treatment, graded according to the NCI CTCAE v3.0 | 4 weeks after completing standard systemic chemotherapy
  The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States